CLINICAL TRIAL: NCT02501226
Title: Effectiveness of the First French Psychoeducational Program on Unipolar Depression: Study Protocol for a Randomized Controlled Trial.
Brief Title: Effectiveness of the First French Psychoeducational Program on Unipolar Depression
Acronym: PURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Groupe Hospitalier de la Rochelle Ré Aunis (Other); Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Général de Béziers (Unknown); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire de Nice (Other); Centre Hospitalier de l'Agglomération de Nevers (Other); Centre Psychothérapique de Nancy (Other); Hôpitaux à Bron (Other); Assistance Publique - Hôpitaux de Paris (Other); Centre Hospitalier Esquirol (Other); Centre Hospitalier Sainte-Marie, Nice (Unknown); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9532
Record Dates: First submitted 2015-07-10; First posted 2015-07-17 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Unipolar Depressed Outpatients; Mild Severity; Without Psychotic Features
Keywords: Psychiatry; Depression; Psychoeducation; Randomized controlled trial; Treatment adherence; Remission
MeSH Terms: conditions — Depression; Treatment Adherence and Compliance | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Treatment as usual
  Interventions: Other: Treatment as usual
- Interventional group (Experimental): ENVIE psychoeducational program
  Interventions: Behavioral: ENVIE psychoeducational program

INTERVENTIONS:
Other: Treatment as usual — Treatment as usual consisting of clinical management including assessment of the psychiatric symptoms and subsequent prescription of antidepressants.
  Arms: Control group
Behavioral: ENVIE psychoeducational program — The intervention will consist of 9 weekly, 90 min sessions led by two animators. The program ENVIE will provide:1.Presentation of the program 2.Education on depressive symptoms. 3.Information about the causes leading to depression. 4.The depression's consequences. 5.Teaching about the last neurobiological and neuroanatomical knowledges about depression, through didactic presentations. 6.How to recognize his own mood state, the prodromal symptoms of relapse. 7.Didactic explanation of the neurobiological action of antidepressant, and other evidence-based medical treatments. 8 and 9. Recommendations about lifestyle and skills of behavioral activation.To enhance the active role of the patient, each session will be accompanied with homework for the patient.
  The sessions may be carried out remotely, by videoconference.
  Arms: Interventional group

SUMMARY:
Background. Major Depressive Disorder (MDD) is highly prevalent and was associated with greater morbidity, mortality (including suicide), and healthcare costs. By 2030, MDD will become the leading cause of disability in high-income countries. Notably, among patients with a previous experience of a major depressive episode, it was indeed estimated that up to 85% of those patients will suffer from relapse. Two main factors were associated with a significantly higher risk of relapse: poor medication adherence and low self-efficacy in disease management. Interestingly, these issues could become the targets of psychoeducational programs for chronic diseases. Indeed psychoeducational program for depression are recommended in international guidelines, but have not yet been proposed in France.

Methods/Design: The investigators propose to evaluate the first French psychoeducational program for depression named "ENVIE" in a multicenter randomized controlled trial. Its aim is to educate patients on the latest knowledge on depression and effective treatments through didactic and interactive sessions. Patients will experiment the latest innovating psychological skills (from acceptance and commitment therapy) to cope with depressive symptoms and maintain motivation in behavioral activation. In total, 332 unipolar non-chronic (< 2 years) outpatients with moderate to severe depression, without psychotic features, will be randomly allocated to the add-on ENVIE program (N=166) or to a waiting list (N=166). The follow-up will last 15 months and include 5 assessment visits (enrollment, 3, 6, 9, 12, 15 months).

Discussion. If the proposed trial shows the effectiveness of the intervention, but also an increased remission rate in depressed outpatients at 15-months post-inclusion, in addition to improved treatment adherence in patients, it will further promotes arguments in favor of a wide dissemination of psychoeducational programs for depression.

DETAILED DESCRIPTION:
The investigators propose to study the rate of remission at 15-month follow-up and time to achieve remission of index episode in a multicentric randomized controlled trial using ENVIE program and treatment as usual versus treatment as usual only. The investigators will include depressed subjects suffering from non a first depressive episode as well as recurrent episode.The eligible patients will be randomized into two groups (computer-generated randomisation in a 1 :1 ratio, blocked in groups of 4, stratified on the number of episodes : 1 , 2 , 3 and more). Only outpatients consulting in the investigation centres will be recruited. Sociodemographic data, psychiatric diagnoses using Mini-International Neuropsychiatric Interview (M.I.N.I.) and Screening Interview for Axis II Disorder (SCID-II) for borderline personality disorder, pharmacological treatment will be also recorded. Patients will be assessed by clinicians blind to treatment allocation, at inclusion (before intervention) and at 3 months (end of the intervention), 6, 9 and 15 months after the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* with a main diagnosis of non-psychotic non-chronic (<2 years) major depressive episode (DSM-IV criteria) of moderate to severe intensity (Montgomery Asberg Depression Scale score > 24)
* taking at least one antidepressant
* able to speak, read and understand French
* and able to give written informed consent

Exclusion Criteria:

* current psychotic features
* duration of current depressive episode >2 years
* current organic mental disorder or mental retardation, or severe comorbid medical condition
* lifetime history of schizophrenia, or schizoaffective or bipolar disorder, manic, hypomanic, or mixed episodes according to DSM-IV criteria
* sensory or cognitive disabilities
* having a relationship or being employed by the sponsor or investigator.
* We will also exclude patients who are planning a long stay outside the region preventing compliance with the scheduled visits, and subjects participating in another trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Rate of remission of index episode at 15-months without relapse during follow-up | 15 months after enrollment
  The primary endpoint will be the remission rate of the index episode at 15 months post-inclusion, defined by a Montgomery and Asberg Depression Rating Scale (MADRS) score ≤ 12 over an 8-week period, and without relapse during follow-up.

SECONDARY OUTCOMES:
Variation of depressive intensity using Medication Adherence Rating Scale (MADRS) | Between enrollment, and 3, 6, 9 and 15 months after enrollment
Evolution of MADRS and BDI scores during follow-up; | At the enrollment, then at 3, 6, 9 and 15 months
Rate of response (decrease of MADRS score by 50%) | At 15 months after enrollment
Rate of relapse (MADRS > 12 after remission of index episode) | At 15 months after enrollment
Rate of hospitalisation during follow-up period | At the enrollment, then at 3, 6, 9 and 15 months
Variation of global functioning using the Functioning Assessment Short Test | Between enrollment, and 9 and 15 months after enrollment
Variation of quality of life using World Health Organization Quality Of Life measure-26 | Between enrollment, and 9 and 15 months after enrollment
Variation of treatment adherence using MADRS | Between enrollment and 15 months after enrollment
Variation of benzodiazepines doses (data collection, no modification treatment according to the protocol) | Between enrollment and 15 months after enrollment
Discontinuation rate of the antidepressant treatment . | At 15 months after enrollment
Variation of depressive intensity using Beck Depression Inventory (BDI) scores | Between enrollment, and 3, 6, 9 and 15 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Emilie OLIE, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

REFERENCES:
- [Derived] Ducasse D, Courtet P, Seneque M, Genty C, Picot MC, Schwan R, Olie E. Effectiveness of the first French psychoeducational program on unipolar depression: study protocol for a randomized controlled trial. BMC Psychiatry. 2015 Nov 17;15:294. doi: 10.1186/s12888-015-0667-7. PMID 26578205